CLINICAL TRIAL: NCT00149292
Title: A Randomized, Double-Blind Comparison of LY2140023, Olanzapine, and Placebo in the Treatment of Patients With Schizophrenia
Brief Title: Study of LY2140023 in Schizophrenia Comparing LY2140023, Olanzapine, and Placebo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Denovo Biopharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9777; H8Y-BD-HBBD
Record Dates: First submitted 2005-09-02; First posted 2005-09-08 (Estimated); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — LY 2140023; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Investigators and patients were blinded to each patient's treatment. Only a pharmacist or designated person at the study site were unblinded to each patient's treatment.

ARMS (3):
- LY2140023 (Experimental): 40 mg LY2140023 BID for 28 days
  Interventions: Drug: LY2140023
- Olanzapine (Active Comparator): 15 mg Olanzapine once daily (QD) for 28 days
  Interventions: Drug: olanzapine
- Placebo (Placebo Comparator): placebo for 28 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: LY2140023
  Arms: LY2140023
Drug: olanzapine
  Arms: Olanzapine
Drug: placebo
  Arms: Placebo

SUMMARY:
Assess the efficacy of a new drug (a receptor agonist that modulates the glutamatergic activity) in the treatment of schizophrenia.

The primary objective of this study is to determine if a mGlu2/3 agonist dosed for 28 days is superior to placebo in the treatment of patients with schizophrenia as measured by the Positive and Negative Symptom Scales (PANSS) total score.

DETAILED DESCRIPTION:
The primary objective of this study was to determine if LY2140023 dosed at 40 mg twice daily (BID) for 28 days was superior to placebo in the treatment of patients with schizophrenia as measured by the Positive and Negative Syndrome Scale (PANSS) total score. The secondary objectives of the study were to assess the safety and tolerability of LY2140023 compared with placebo and olanzapine; efficacy of LY2140023 compared with placebo in change from baseline to Visit 8 in the PANSS positive symptom subset score; efficacy of LY2140023 compared with placebo in the responder rate (defined as 25% or more decrease from baseline to Visit 8) in the PANSS total score; efficacy of LY2140023 compared with placebo in responder rate (defined as 25% or more decrease from baseline to Visit 8) in the PANSS positive symptom subset score; efficacy of LY2140023 compared with placebo in change from baseline to Visit 8 in the PANSS negative symptom subset score; efficacy of LY2140023 compared with placebo in change from baseline to Visit 8 in mood and anxiety as measured by the Hamilton Anxiety Scale (HAMA) total score; efficacy of LY2140023 compared with placebo in change from baseline to Visit 8 in the Clinical Global Impression-Severity (CGI-S); effect of LY2140023 on prolactin levels of the patients after 4 weeks of treatment; efficacy of olanzapine compared with placebo on the PANSS total score; pharmacokinetics of LY2140023 and LY404039 in patients, and to explore the relationship between exposure and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* meet the DSM-IV criteria for schizophrenia as confirmed by modified SCID

Exclusion Criteria:

* meet the full syndromal criteria for other Axis I disorder
* have taken any depot antipsychotic within 4 weeks before screening
* are taking mood-stabilizing agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2005-08-23 (Actual); Primary Completion 2006-07-17 (Actual); Study Completion 2006-07-17 (Actual)

PRIMARY OUTCOMES:
To determine if a mGlu2/3 agonist (LY2140023) dosed for 28 days is superior to placebo in the treatment of patients with schizophrenia as measured by the Positive and Negative Symptom Scales (PANSS) total score | 28 days
  The primary objective of this study was to determine if LY2140023 dosed at 40 mg twice daily (BID) for 28 days was superior to placebo in the treatment of patients with schizophrenia as measured by the Positive and Negative Symptom Scale (PANSS) total score.

SECONDARY OUTCOMES:
Safety and tolerability of LY2140023 compared with placebo and olanzapine | 28 days
  Safety parameters evaluated included physical and neurological examinations, vital signs, body weight, 12-lead electrocardiograms (ECGs), clinical laboratory tests, prolactin levels, and the record of symptoms. Other safety measures included the Barnes Akathisia Scale (BAS), Simpson- Angus Scale (SAS), and the Abnormal Involuntary Movement Scale (AIMS).
Efficacy of LY2140023 compared with placebo in change from baseline to Visit 8 in the PANSS positive symptom subset score | 28 days
  The secondary efficacy variables include the change from baseline in the PANSS positive symptoms subset score, the PANSS negative symptom subset score, CGI-S score, and HAMA total score. A patient will be included in the analysis if he or she has a baseline and at least one post-baseline measure.
Efficacy of LY2140023 compared with placebo in the responder rate in the PANSS total score | 28 days
  Efficacy of LY2140023 compared with placebo in the responder rate (defined as 25% or more decrease from baseline to Visit 8) in the PANSS total score
Efficacy of LY2140023 compared with placebo in responder rate in the PANSS positive and negative symptom subset score | 28 days
  Efficacy of LY2140023 compared with placebo in responder rate (defined as 25% or more decrease from baseline to Visit 8) in the PANSS positive and negative symptom subset score

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM-5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Russia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Village Nikolskoe

REFERENCES:
- [Derived] Kinon BJ, Millen BA, Zhang L, McKinzie DL. Exploratory analysis for a targeted patient population responsive to the metabotropic glutamate 2/3 receptor agonist pomaglumetad methionil in schizophrenia. Biol Psychiatry. 2015 Dec 1;78(11):754-62. doi: 10.1016/j.biopsych.2015.03.016. Epub 2015 Mar 19. PMID 25890643